CLINICAL TRIAL: NCT06515106
Title: Antibody-mediated LGI1 Encephalitis: Symptoms, Biomarkers, and Mechanisms of the Chronic Phase of the Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PI23/00858
Record Dates: First submitted 2024-03-26; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Limbic Encephalitis With LGI1 Antibodies
Keywords: Cognitive Impairment; Encephalitis; Autoimmune; Cognitive rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Encephalitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antibody-mediated LGI1 encephalitis patients (Experimental): Participants of a prospective cohort in post-acute phase of the Antibody-mediated NMDA Receptor Encephalitis that will received a behavioral treatment.
  Interventions: Behavioral: Remote cognitive rehabilitation program

INTERVENTIONS:
Behavioral: Remote cognitive rehabilitation program — Behavioral: Remote cognitive rehabilitation program Remote cognitive rehabilitation program will be performed through an online validated platform (Guttmann NeuroPersonalTrainer: https://gnpt.es/) run by the psychologists team. This is a Sanitary Product with CE certification (Sanitary Product RPS/430/2014; International Patent [PCT/ES2008/00677]) and here will be used within its approved indications. The rehabilitation program will increase in difficulty and decrease in frequency during the first year of follow-up (V1-V3).

SUMMARY:
The encephalitis mediated by antibodies against Leucine-rich, glioma inactivated 1 protein (anti-LGI1 encephalitis) predominantly affects men (M:F, 6:4) and mostly older than 60 years. The disease has two distinct clinical phases: The acute phase in which the majority of patients develop severe short-term memory deficits (unable to remember events or experiences that occurred a few minutes earlier). This memory impairment can be preceded or accompanied by one or more of the following: hyponatremia (60% of patients), a highly distinctive type of seizures called facio-brachial dystonic seizures (~40% of patients), along with confusion, irritability and other types of focal seizures or less frequently, generalized seizures. In addition, many patients at this stage have symptoms of REM sleep behavior disorder. In this stage, the CSF may show pleocytosis or mild increase of proteins, the EEG is usually abnormal, and in ~60% of the patients the MRI shows typical increased FLAIR signal in medial temporal lobes (11). There is a clinical sub-phenotype (~13% of patients) in which the disease presents as a rapidly progressive cognitive decline without the indicated FLAIR MRI changes. About 70% of patients improve rapidly with corticosteroids and immunotherapy (eg, intravenous immunoglobulins and/or plasma exchange), but the improvement is often partial. After the acute phase, there is a chronic or residual phase which represents the interval from improvement of initial symptoms until the disease is considered no longer active and the remaining symptoms are thought to be irreversible. This chronic phase may take several months (it has been less well studied), and is characterized by the absence of CSF pleocytosis and inflammatory MRI changes (albeit this may show residual hippocampal atrophy), and very low or undetectable titers of serum antibodies. Most patients are unable to return to their job or previous activities due to residual (irreversible) memory or cognitive deficits accompanied by signs of moderate brain atrophy. In addition, we and others have shown that about 27-35% of patients have relapsing symptoms after improving from the acute phase (. Although acute symptomatic seizures (facio-brachial dystonic and others) occur in ~90% of patients during the acute phase of the disease, less than 10% of patients develop chronic epilepsy often associated with hippocampal sclerosis. Therefore, the prevailing concept on this disease suggests a syndrome and clinical course in which the acute phase shows rapid, albeit partial, response to immunotherapy, and the symptoms of the chronic phase represent a burnout or irreversible process, in which the disease is no longer active, and the potential improvement of remaining symptoms is uncertain.

Here investigators postulate that a better knowledge of this stage will improve treatment decisions and outcome.

In Aim 1, the post-acute stage will be clinically characterized.

In Aim 2, the impact of cognitive rehabilitation will be assessed.

In Aim 3, a mouse model of anti-LGI1 encephalitis will be used to determine the underlying mechanisms and treatment of the postacute stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Antibody-mediated LGI-1 encephalitis in the post-acute stage of the disease;
* Patients has been discharged from hospital (acute phase).

Exclusion Criteria:

* Inability to obtain informed consent;
* Inability to travel to the center.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Age | 12 months
  Age measured in years
Gender | 12 months
  Male or female
Handedness | 12 months
  Right- or Left-handed
General medical history | 12 months
  Description of the most important issues compiled in the general medical history of the participant
Allergies | 12 months
  List of allergies of each participant
Symptoms related to anti-LGI1 encephalitis | 12 months
  Detailed description of symptoms experienced before, during and after the post-acute phase of anti-LGI1 encephalitis.
Treatments | 12 months
  All treatments in which the participant is being involved.
Functional status | 12 months
  Functional status according to Modified Rankin Scale (mRS).
  Modified Rankin Scale:
  - Range: from 0 points (no symptoms) to 6 points (dead).
Intelligence Quotient | 12 months
  Estimated through General Ability Index (GAI; from Weschler Adult Intelligence Scale - IV (WAIS-IV).
  This index is obtained through Verbal Comprehension Index (VCI) and Perceptual Reasoning Index (PRI).
  Range of GAI: from 40 to 160. Higher is better. Range of VCI: from 50 to 150. Higher is better. Range of PRI: from 50 to 150. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal working memory | 12 months
  Verbal Working Memory: Working Memory Index (WMI) from WAIS-IV.
  - Range of WMI: from 50 to 150. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Phonological loop | 12 months
  Assessed by Forward order span of Digit span subtest from WAIS-IV.
  - Range: from 0 to 9
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual working memory | 12 months
  Visual Working Memory: Spatial location subtest from Weschler Memory Scale - IV (WMS-IV).
  - Range of Spatial Location subtest: from 0 to 32. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal learning | 12 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC
  - Total learning: range: from 0 to 80. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Proactive interference verbal memory | 12 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC).
  - Interference list: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Short-term verbal memory | 12 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC).
  - Short-term memory free recall: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Long-term verbal memory | 12 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC):
  - Long-term memory free recall: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal recognition memory | 12 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC).
  - Word-list Recognition: range: 0 to 15. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal discrimination memory | 12 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC)
  Discrimination index of word-list: False positives + omissions of recognition between 44 total words to recognize. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Verbal retention memory | 12 months
  Assessed by:
  Adults: España - Complutense Auditory-Verbal Learning Test (Test de Aprendizaje Verbal España - Complutense; TAVEC); or Infants: España - Complutense Auditory-Verbal Learning Test for Children (Test de Aprendizaje Verbal España - Complutense Infantil; TAVECI)
  - Retention index: percentatge of Long-term memory free recall between Short-term memory free recall. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Immediate visual memory | 12 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Immediate visual memory: range: from 0 to 36. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Delayed visual memory | 12 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Delayed visual memory: range: from 0 to 12. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual retention memory | 12 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Retention index: percentatge of Long-term memory free recall between the Higher punctuation at Trial 2 or 3. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual recognition memory | 12 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Figure Recognition: range: from 0 to 6. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visual discrimination memory | 12 months
  Assessed by: Brief Visuospatial Memory Test - Revised (BVMT-R)
  - Discrimination index: figure recognized minus false positives. Range: from -6 to 6. Higher is better.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Processing speed | 12 months
  Symbol Search subtest (WAIS-IV)
  - Total (correct answers less incorrect answers): from 0 to 60
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
TMT-A | 12 months
  Trail Making Test part A (TMT-A):
  - Time in seconds: from 0 to infinity.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Naming | 12 months
  Assessed by: Boston Naming Test (BNT)
  - Total correct: from 0 to 60
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Naming with cues | 12 months
  Assessed by: Boston Naming Test (BNT)
  - Total correct with phonemic cue: from 0 to 60
Latency in naming | 12 months
  Assessed by: Boston Naming Test (BNT)
  - Time to complete test in seconds
Semantic fluency | 12 months
  Number of name of animals recalled in 1 minute: range: from 0 to infinity.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Phonemic fluency | 12 months
  Number of words started by letter "M" recalled in 1 minute:
  - Range: from 0 to infinity.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Visuospatial skills | 12 months
  Number location subtest of the Visual-Object Spatial and Perceptual battery.
  - Range: from 0 to 10
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Symbolic gesture right hand - order | 12 months
  Symbolic gesture right hand - order subtest from Test Barcelona - Revised
  - Range: from 0 to 10
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Symbolic gesture left hand - order | 12 months
  Symbolic gesture left hand - order subtest from Test Barcelona - Revised
  - Range: from 0 to 10
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Symbolic gesture right hand - imitation | 12 months
  Symbolic gesture right hand - imitation subtest from Test Barcelona
  - Range: from 0 to 10
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Symbolic gesture left hand - imitation | 12 months
  Symbolic gesture left hand - imitation subtest from Test Barcelona - Revised
  - Range: from 0 to 10
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Bilateral ideomotor praxis - imitation | 12 months
  Bilateral ideomotor praxis imitation subtest from Test Barcelona
  - Range: from 0 to 10
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Stroop test - word subtest | 12 months
  - Words: words read in 45 seconds
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Stroop test - color subtest | 12 months
  - Colour: colours distinguished in 45 seconds.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Stroop test - word-color subtest | 12 months
  - Word-colour: colours distinguished in 45 seconds.
  Raw scores were transformed into standard T-scores (mean 50 ± standard deviation [SD] 10) and a score below 35 (≤ 1.5 SD below normative mean, or the equivalent ≤9th percentile) was considered significantly decreased.
Prensence of psychiatric symptoms or disorders | 12 months
  Number of participants with psychiatric symptoms/disorders following DSM-IV-TR guidelines (psychotic symptoms, symptoms of depression, symptoms of mania, global functioning).
Sleep microstructure - Total study time | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Total sleep time: minutes
Sleep microstructure - Total sleep time | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Total sleep time: minutes
Sleep microstructure - Sleep efficiency | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Sleep efficiency: based on total study time and total sleep time
Sleep microstructure - Time to sleep onset | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time to sleep onset: minutes
Sleep microstructure - Time in stage N1 | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage N1: minutes
Sleep microstructure - Time in stage N2 | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage N2: minutes
Sleep microstructure - Time in stage N3 | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage N3: minutes
Sleep microstructure - Time in stage R | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Time in stage R: minutes
Sleep microstructure - First epoch of N1 | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of N1: minutes
Sleep microstructure - First epoch of N2 | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of N2: minutes
Sleep microstructure - First epoch of N3 | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of N3: minutes
Sleep microstructure - First epoch of REM | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - First epoch of REM: minutes
Sleep microstructure - REM/NREM time ratio | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - REM/NREM time ratio
Sleep microstructure - Number of arousals | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Number of arousals (total)
Sleep microstructure - Arousal Index | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Arousal Index
Sleep microstructure - Confusional arousals | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Confusional arousals: Yes or No
Sleep microstructure - Direct transition from N3 to W | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Direct transition from N3 to W: yes or no
Sleep microstructure - Delta arousals | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Delta arousals: yes, no or unknown
Sleep microstructure - Wake after sleep | 12 months
  It will be adapted to patient's sleep habits (~23:00 to 07:30) using a digital polygraph (Deltamed). This includes EEG in 43 scalp channels + 11 channels for electrooculography, electrocardiography, electromyography, and audiovisual recording (sampling rate 256 Hz). Sleep stages will be scored manually (AASM criteria) using 30-s epochs, with modifications depending on sleep alterations, as reported.
  Parameters:
  - Wake after sleep: hour
Adherence to cognitive treatment - 6 months | 6 months
  Percentage of sessions performed in 6 months out of 48 (sessions performed out of 48 x 100)
Adherence to cognitive treatment - 9 months | 9 months
  Percentage of sessions performed in 9 months (sessions performed out of 54 x 100)
Adherence to cognitive treatment - 12 months | 12 months
  Percentage of sessions performed in 9 months out of 60 (sessions performed out of 60 x 100)
Cardiovagal evaluation. (Composite autonomic scoring scale) | 12 months
  Continuous electrocardiogram heart rate changes during deep breathing and postural changes (beats per minute).Composite autonomic scoring scale minimun 0, maximum 3, higher scores mean a worse outcome.
Valsava ratio | 12 months
  Continuous electrocardiogram heart rate changes during Valsalva manoeuvre (ratio).
Sympathetic evaluation (Composite autonomic scoring scale) | 12 months
  Beat-to-beat blood pressure changes to isometric exercise, Valsalva manoeuvre and postural changes, (mmHg). Composite autonomic scoring scale minimun 0, maximum 4, higher scores mean a worse outcome
Composite Autonomic Symptom Score (Compass-31) | 12 months
  Self-scoring Compass 31 autonomic assessment. Minimum 0, maximum 100, higher scores mean a worse outcome.
Electromyography (EMG) | 12 months
  Needle recording electrode will be inserted into different muscles (orbicularis oris, extensor indicis propius, tibialis anterior).Presence of abnormal discharges will be recorded (0 none to 4 maximum).
Brainstem reflex | 12 months
  Trigeminal blink reflex, mediated by trigemino-facial ponto-medullary -circuits will be assessed. Surface recording electrodes will be attached over the orbicularis oculi in both sides with active electrode over the middle part of the lower eyelid and the reference at the lateral cantus of the eye . Stimulating electrodes will be placed over the supraorbital nerve. Ipsilateral (R1, R2) and contralateral responses (R2c) latencies measured in ms will be analyzed
MRI | 12 months
  It will be conducted on a 3 Tesla Prisma scanner using a 32-channel head coil. Scanning takes ~50 min including 3D T1-weighted in sagittal plane; T2*axial EPI; axial diffusion weighted EPI; 3D sagittal FLAIR; resting state functional MRI and glutamate and H2O univoxel spectroscopy in dorsolateral prefrontal cortex and hippocampus. There is no contrast used for the MRI scans
  Outcome for MRI is normal or abnormal. Investigators will review all MRI sequences and determine if the MRI is abnormal and then describe the abnormality or abnormalities seen.
EEG: normalcy | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  - Normalcy: yes or no.
EEG: time awake | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Time awake: percentage
EEG: time in drowsiness | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Time in drowsiness: percentage
EEG: time asleep | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Time asleep: percentage
EEG: epileptiform activity | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Epileptiform activity: yes or no
EEG: seizures | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Seizures: yes or no
EEG: slowing | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - EEG slowing: yes or no
EEG: Changes with Intermittent Light Stimulation | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Changes with Intermittent Light Stimulation: yes or no
EEG: Changes with hyperventilation | 12 months
  It will include standard clinical EEG protocol (43 channels, 512 Hz18) (primary variables), and EEG reactivations of memories prior to new trials (secondary variables) while participants perform WM tasks, which will be synchronized with the task software in a laptop. The memory content from alpha power across electrodes will be related to the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Performances of the subjects produces a reactivation of memory prior to new trials while participants perform working memory tasks, and relate the decoding accuracy in different task periods to disease treatment and recovery and to behavioral parameters (WM precision, serial biases).
  Parameters:
  - Changes with hyperventilation: yes or no

SECONDARY OUTCOMES:
LGI-1 antibodies | 12 months
  Determined with brain tissue immunohistochemistry and cell - based assays
HLA genotyping | 12 months
  performed by standard techniques based on DNA - PCR and polymorphism identification by reverse hybridization with specific probes and fluorescence labelling of hybridized fragments (PCR - SSOP) (Immucor GTI Diagnostics Inc.Waukesha USA) in combination with genomic DNA sequencing by Sanger methodology (PCRSBT).
Immune/inflammatory signaling-target gene expression pathways | 12 months
  RNA/NanoString analysis of targeted gene expression related to activation/function of B cells, T cells, microglia, and other interleukin/ chemokine signaling. Whole blood/CSF will be collected using PAXgene® Blood RNA tubes (Qiagen) shipped to the centers. Total RNA will be extracted using PAXgene® Blood RNA Kit (Qiagen). RNA samples are quantified using Qubit 2.0 Fluorometer (Life Technologies) and RNA integrity is determined with Agilent 2100 Bioanalyzer (Agilent Technologies). Expression levels of 44 genes related to immunological pathways and cytokines (Annex,Table) will be measured with the nCounter® Digital Analyzer (NanoString), as reported (Armangue et al., Mol Genet Metab 2017;122:134-9). Twenty healthy participants will serve as controls (single evaluation).
NfL levels | 12 months
  determined in serum and CSF using the SiMoA Quanterix technique, as reported (Guasp et al., Neurology 2022;98:e1489 - 98). Age-and sex-matched healthy participants from previous studies will serve as controls.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Dalmau, MD, PhD, Principal Investigator — Hospital Clínic; Lorena Rami, PhD, Principal Investigator — Fundacion Clinic per a la Recerca Biomédica
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Dalmau J, Graus F. Antibody-Mediated Encephalitis. N Engl J Med. 2018 Mar 1;378(9):840-851. doi: 10.1056/NEJMra1708712. No abstract available. PMID 29490181
- [Background] Dalmau J, Geis C, Graus F. Autoantibodies to Synaptic Receptors and Neuronal Cell Surface Proteins in Autoimmune Diseases of the Central Nervous System. Physiol Rev. 2017 Apr;97(2):839-887. doi: 10.1152/physrev.00010.2016. PMID 28298428
- [Background] Hughes EG, Peng X, Gleichman AJ, Lai M, Zhou L, Tsou R, Parsons TD, Lynch DR, Dalmau J, Balice-Gordon RJ. Cellular and synaptic mechanisms of anti-NMDA receptor encephalitis. J Neurosci. 2010 Apr 28;30(17):5866-75. doi: 10.1523/JNEUROSCI.0167-10.2010. PMID 20427647
- [Background] Planaguma J, Leypoldt F, Mannara F, Gutierrez-Cuesta J, Martin-Garcia E, Aguilar E, Titulaer MJ, Petit-Pedrol M, Jain A, Balice-Gordon R, Lakadamyali M, Graus F, Maldonado R, Dalmau J. Human N-methyl D-aspartate receptor antibodies alter memory and behaviour in mice. Brain. 2015 Jan;138(Pt 1):94-109. doi: 10.1093/brain/awu310. Epub 2014 Nov 11. PMID 25392198
- [Background] Petit-Pedrol M, Sell J, Planaguma J, Mannara F, Radosevic M, Haselmann H, Ceanga M, Sabater L, Spatola M, Soto D, Gasull X, Dalmau J, Geis C. LGI1 antibodies alter Kv1.1 and AMPA receptors changing synaptic excitability, plasticity and memory. Brain. 2018 Nov 1;141(11):3144-3159. doi: 10.1093/brain/awy253. PMID 30346486
- [Background] Titulaer MJ, McCracken L, Gabilondo I, Armangue T, Glaser C, Iizuka T, Honig LS, Benseler SM, Kawachi I, Martinez-Hernandez E, Aguilar E, Gresa-Arribas N, Ryan-Florance N, Torrents A, Saiz A, Rosenfeld MR, Balice-Gordon R, Graus F, Dalmau J. Treatment and prognostic factors for long-term outcome in patients with anti-NMDA receptor encephalitis: an observational cohort study. Lancet Neurol. 2013 Feb;12(2):157-65. doi: 10.1016/S1474-4422(12)70310-1. Epub 2013 Jan 3. PMID 23290630
- [Background] Granerod J, Ambrose HE, Davies NW, Clewley JP, Walsh AL, Morgan D, Cunningham R, Zuckerman M, Mutton KJ, Solomon T, Ward KN, Lunn MP, Irani SR, Vincent A, Brown DW, Crowcroft NS; UK Health Protection Agency (HPA) Aetiology of Encephalitis Study Group. Causes of encephalitis and differences in their clinical presentations in England: a multicentre, population-based prospective study. Lancet Infect Dis. 2010 Dec;10(12):835-44. doi: 10.1016/S1473-3099(10)70222-X. Epub 2010 Oct 15. PMID 20952256
- [Background] van Sonderen A, Petit-Pedrol M, Dalmau J, Titulaer MJ. The value of LGI1, Caspr2 and voltage-gated potassium channel antibodies in encephalitis. Nat Rev Neurol. 2017 May;13(5):290-301. doi: 10.1038/nrneurol.2017.43. Epub 2017 Apr 18. PMID 28418022
- [Background] Gable MS, Sheriff H, Dalmau J, Tilley DH, Glaser CA. The frequency of autoimmune N-methyl-D-aspartate receptor encephalitis surpasses that of individual viral etiologies in young individuals enrolled in the California Encephalitis Project. Clin Infect Dis. 2012 Apr;54(7):899-904. doi: 10.1093/cid/cir1038. Epub 2012 Jan 26. PMID 22281844
- [Background] Armangue T, Spatola M, Vlagea A, Mattozzi S, Carceles-Cordon M, Martinez-Heras E, Llufriu S, Muchart J, Erro ME, Abraira L, Moris G, Monros-Gimenez L, Corral-Corral I, Montejo C, Toledo M, Bataller L, Secondi G, Arino H, Martinez-Hernandez E, Juan M, Marcos MA, Alsina L, Saiz A, Rosenfeld MR, Graus F, Dalmau J; Spanish Herpes Simplex Encephalitis Study Group. Frequency, symptoms, risk factors, and outcomes of autoimmune encephalitis after herpes simplex encephalitis: a prospective observational study and retrospective analysis. Lancet Neurol. 2018 Sep;17(9):760-772. doi: 10.1016/S1474-4422(18)30244-8. Epub 2018 Jul 23. PMID 30049614
- [Background] Lai M, Huijbers MG, Lancaster E, Graus F, Bataller L, Balice-Gordon R, Cowell JK, Dalmau J. Investigation of LGI1 as the antigen in limbic encephalitis previously attributed to potassium channels: a case series. Lancet Neurol. 2010 Aug;9(8):776-85. doi: 10.1016/S1474-4422(10)70137-X. Epub 2010 Jun 28. PMID 20580615
- [Background] Irani SR, Alexander S, Waters P, Kleopa KA, Pettingill P, Zuliani L, Peles E, Buckley C, Lang B, Vincent A. Antibodies to Kv1 potassium channel-complex proteins leucine-rich, glioma inactivated 1 protein and contactin-associated protein-2 in limbic encephalitis, Morvan's syndrome and acquired neuromyotonia. Brain. 2010 Sep;133(9):2734-48. doi: 10.1093/brain/awq213. Epub 2010 Jul 27. PMID 20663977
- [Background] Munoz-Sanchez G, Planaguma J, Naranjo L, Couso R, Sabater L, Guasp M, Martinez-Hernandez E, Graus F, Dalmau J, Ruiz-Garcia R. The diagnosis of anti-LGI1 encephalitis varies with the type of immunodetection assay and sample examined. Front Immunol. 2022 Dec 15;13:1069368. doi: 10.3389/fimmu.2022.1069368. eCollection 2022. PMID 36591253
- [Background] van Sonderen A, Thijs RD, Coenders EC, Jiskoot LC, Sanchez E, de Bruijn MA, van Coevorden-Hameete MH, Wirtz PW, Schreurs MW, Sillevis Smitt PA, Titulaer MJ. Anti-LGI1 encephalitis: Clinical syndrome and long-term follow-up. Neurology. 2016 Oct 4;87(14):1449-1456. doi: 10.1212/WNL.0000000000003173. Epub 2016 Sep 2. PMID 27590293
- [Background] Arino H, Armangue T, Petit-Pedrol M, Sabater L, Martinez-Hernandez E, Hara M, Lancaster E, Saiz A, Dalmau J, Graus F. Anti-LGI1-associated cognitive impairment: Presentation and long-term outcome. Neurology. 2016 Aug 23;87(8):759-65. doi: 10.1212/WNL.0000000000003009. Epub 2016 Jul 27. PMID 27466467
- [Background] Iranzo A, Graus F, Clover L, Morera J, Bruna J, Vilar C, Martinez-Rodriguez JE, Vincent A, Santamaria J. Rapid eye movement sleep behavior disorder and potassium channel antibody-associated limbic encephalitis. Ann Neurol. 2006 Jan;59(1):178-81. doi: 10.1002/ana.20693. PMID 16278841
- [Background] de Bruijn MAAM, van Sonderen A, van Coevorden-Hameete MH, Bastiaansen AEM, Schreurs MWJ, Rouhl RPW, van Donselaar CA, Majoie MHJM, Neuteboom RF, Sillevis Smitt PAE, Thijs RD, Titulaer MJ. Evaluation of seizure treatment in anti-LGI1, anti-NMDAR, and anti-GABABR encephalitis. Neurology. 2019 May 7;92(19):e2185-e2196. doi: 10.1212/WNL.0000000000007475. Epub 2019 Apr 12. PMID 30979857
- [Background] Ramberger M, Berretta A, Tan JMM, Sun B, Michael S, Yeo T, Theorell J, Bashford-Rogers R, Paneva S, O'Dowd V, Dedi N, Topia S, Griffin R, Ramirez-Franco J, El Far O, Baulac S, Leite MI, Sen A, Jeans A, McMillan D, Marshall D, Anthony D, Lightwood D, Waters P, Irani SR. Distinctive binding properties of human monoclonal LGI1 autoantibodies determine pathogenic mechanisms. Brain. 2020 Jun 1;143(6):1731-1745. doi: 10.1093/brain/awaa104. PMID 32437528
- [Background] Ohkawa T, Fukata Y, Yamasaki M, Miyazaki T, Yokoi N, Takashima H, Watanabe M, Watanabe O, Fukata M. Autoantibodies to epilepsy-related LGI1 in limbic encephalitis neutralize LGI1-ADAM22 interaction and reduce synaptic AMPA receptors. J Neurosci. 2013 Nov 13;33(46):18161-74. doi: 10.1523/JNEUROSCI.3506-13.2013. PMID 24227725
- [Background] Guasp M, Rosa-Justicia M, Munoz-Lopetegi A, Martinez-Hernandez E, Armangue T, Sugranyes G, Stein H, Borras R, Prades L, Arino H, Planaguma J, De-La-Serna E, Escudero D, Llufriu S, Sanchez-Valle R, Santamaria J, Compte A, Castro-Fornieles J, Dalmau J; Spanish anti-NMDAR Encephalitis Study Group. Clinical characterisation of patients in the post-acute stage of anti-NMDA receptor encephalitis: a prospective cohort study and comparison with patients with schizophrenia spectrum disorders. Lancet Neurol. 2022 Oct;21(10):899-910. doi: 10.1016/S1474-4422(22)00299-X. PMID 36115362
- [Background] Irani SR, Stagg CJ, Schott JM, Rosenthal CR, Schneider SA, Pettingill P, Pettingill R, Waters P, Thomas A, Voets NL, Cardoso MJ, Cash DM, Manning EN, Lang B, Smith SJ, Vincent A, Johnson MR. Faciobrachial dystonic seizures: the influence of immunotherapy on seizure control and prevention of cognitive impairment in a broadening phenotype. Brain. 2013 Oct;136(Pt 10):3151-62. doi: 10.1093/brain/awt212. Epub 2013 Sep 6. PMID 24014519
- [Background] Diaz Baquero AA, Franco-Martin MA, Parra Vidales E, Toribio-Guzman JM, Bueno-Aguado Y, Martinez Abad F, Perea Bartolome MV, Asl AM, van der Roest HG. The Effectiveness of GRADIOR: A Neuropsychological Rehabilitation Program for People with Mild Cognitive Impairment and Mild Dementia. Results of a Randomized Controlled Trial After 4 and 12 Months of Treatment. J Alzheimers Dis. 2022;86(2):711-727. doi: 10.3233/JAD-215350. PMID 35124649

DOCUMENTS (2):
  • Study Protocol (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT06515106/Prot_000.pdf
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT06515106/ICF_001.pdf